CLINICAL TRIAL: NCT06709079
Title: Study on the Effect and Mechanism of Aescine Sodium in the Treatment of Allergic Rhinitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cheng Lei (Other)
Responsible Party: Sponsor-Investigator, Cheng Lei, chief physician, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-SR-796
Record Dates: First submitted 2024-01-21; First posted 2024-11-29 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allergic rhinitis (Experimental): Preoperatively, patients with AR were given 2 tablets of Aescine Sodium Tablets (Ocai®, Green Leaf Pharmaceuticals) to be taken after meals, once in the morning and once in the evening, for a period of 20 days.
  Interventions: Drug: Aescine Sodium Tablets (Ocai®, Green Leaf Pharmaceuticals)

INTERVENTIONS:
Drug: Aescine Sodium Tablets (Ocai®, Green Leaf Pharmaceuticals) — Preoperatively, patients with AR were given 2 tablets of Aescine Sodium Tablets (Ocai®, Green Leaf Pharmaceuticals) to be taken after meals, once in the morning and once in the evening, for a period of 20 days.

SUMMARY:
Allergic rhinitis is a common chronic non-infectious inflammatory disease of the upper respiratory tract, which affects patients' health, quality of life and work efficiency for a long time. Clinical manifestations are mainly nasal congestion, paroxysmal sneezing, clear watery nasal discharge and nasal itching, among which nasal congestion caused by nasal mucosal edema is the main manifestation of allergic rhinitis. Nasal mucosa has a rich network of arteriovenous anastomosis, and there are many large venous sinuses constitute a spongy structure, with a strong capacity for expansion and contraction, in the onset of allergic rhinitis, the volume of venous sinuses in the nasal mucosa can be rapidly changed, venous sinus expansion and filling can be induced by nasal mucosal congestion and nasal mucosal edema nasal congestion symptoms. Aescine sodium has been widely used in the clinical treatment of local tissue edema and the effect is remarkable, a large number of clinical results have proved that it has a significant anti-inflammatory, anti-edema, enhance the venous tension, improve blood circulation and anti-allergic effect, can be improved through the improvement of the vascular endothelial cell barrier, and enhance the epithelial cells close connection to improve the local edema and acute inflammation. The current treatment strategies for allergic rhinitis mainly include environmental control, medication, immunotherapy and health education, however, some patients are still unable to effectively control their symptoms in the long term after standardized treatment, and nasal congestion and runny nose cause great disturbance to the quality of their daily life. Therefore, it is urgent to investigate the mechanism of aescine sodium in relieving nasal mucosal edema in allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-65 years).
* Patients with allergic rhinitis were diagnosed based on clinical history and positive sensitization tests (skin prick test and/or specific IgE).

Exclusion Criteria:

* Received glucocorticoids, immunomodulatory, antihistamine drugs, and other medications that may affect the study results within the last 1 month.
* Nasal diseases such as upper respiratory tract infections, chronic sinusitis with or without nasal polyps, and nasal sinus tumors.
* History of nasal sinus surgery.
* With other immune and allergic diseases.
* Patients with a combination of severe cardiac, cerebrovascular or pulmonary - diseases, aspirin triad, primary ciliary dyskinesia, immune deficiency, and coagulation disorders.
* Pregnant women.
* Smokers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Rhinoconjunctivitis Quality of Life Questionnaire | baseline and 20 days
  To measure the functional impairments that are most troublesome to adult patients as a result of their rhinoconjunctivitis. Patients were scored by questionnaire before and after treatment, and the change in score before and after treatment was the primary outcome measure. 7-point scale (0 = not impaired at all - 6 = severely impaired). Higher scores reflect lower quality of life.
Visual analogue scale | baseline and 20 days
  Results Visual analogue scale(VAS) are well validated for the measurement of AR symptoms and correlate well with the ARIA (allergic rhinitis and its impact on asthma) severity classification. Patients were scored by questionnaire before and after treatment, and the change in score before and after treatment was the primary outcome measure.
  Range: 0-10. Higher scores reflect more pain and severity.
The concentration of interleukin 4(IL-4), interleukin 5(IL-5), interleukin 13(IL-13) | baseline and 20 days
  It reflects Th2 immune response in patients with allergic rhinitis.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Al-Digheari A, Mahboub B, Tarraf H, Yucel T, Annesi-Maesano I, Doble A, Lahlou A, Tariq L, Aziz F, El Hasnaoui A. The clinical burden of allergic rhinitis in five Middle Eastern countries: results of the SNAPSHOT program. Allergy Asthma Clin Immunol. 2018 Nov 19;14:63. doi: 10.1186/s13223-018-0298-x. eCollection 2018. PMID 30473712
- [Background] Cheng L, Chen J, Fu Q, He S, Li H, Liu Z, Tan G, Tao Z, Wang D, Wen W, Xu R, Xu Y, Yang Q, Zhang C, Zhang G, Zhang R, Zhang Y, Zhou B, Zhu D, Chen L, Cui X, Deng Y, Guo Z, Huang Z, Huang Z, Li H, Li J, Li W, Li Y, Xi L, Lou H, Lu M, Ouyang Y, Shi W, Tao X, Tian H, Wang C, Wang M, Wang N, Wang X, Xie H, Yu S, Zhao R, Zheng M, Zhou H, Zhu L, Zhang L. Chinese Society of Allergy Guidelines for Diagnosis and Treatment of Allergic Rhinitis. Allergy Asthma Immunol Res. 2018 Jul;10(4):300-353. doi: 10.4168/aair.2018.10.4.300. PMID 29949830
- [Background] Lee HC, Yu HP, Liao CC, Chou AH, Liu FC. Escin protects against acetaminophen-induced liver injury in mice via attenuating inflammatory response and inhibiting ERK signaling pathway. Am J Transl Res. 2019 Aug 15;11(8):5170-5182. eCollection 2019. PMID 31497232
- [Background] Lindner I, Meier C, Url A, Unger H, Grassauer A, Prieschl-Grassauer E, Doerfler P. Beta-escin has potent anti-allergic efficacy and reduces allergic airway inflammation. BMC Immunol. 2010 May 21;11:24. doi: 10.1186/1471-2172-11-24. PMID 20487574
- [Background] Gallelli L. Escin: a review of its anti-edematous, anti-inflammatory, and venotonic properties. Drug Des Devel Ther. 2019 Sep 27;13:3425-3437. doi: 10.2147/DDDT.S207720. eCollection 2019. PMID 31631970